CLINICAL TRIAL: NCT02380079
Title: Part A: Phase IB, Single Site, Dose-Escalation of SCD-101 and Part B: Randomized, Double-Blind, Placebo-Controlled Crossover of SCD-101 in Adults With Homozygous Sickle Cell Disease or S/Beta 0 Thalassemia.
Brief Title: Dose-Escalation Study of SCD-101 in Sickle Cell Disease
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Invenux, LLC (Industry)
Collaborators: State University of New York - Downstate Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: INVX-SCD-101-11
Record Dates: First submitted 2015-02-23; First posted 2015-03-05 (Estimated); Last update posted 2023-03-21 (Actual); Status verified 2023-03

CONDITIONS: Sickle Cell Disease; Sickle-Beta Zero Thalassemia
Keywords: Homozygous Sickle Cell Disease S/Beta 0 Thalassemia
MeSH Terms: conditions — Anemia, Sickle Cell

STUDY DESIGN:
Intervention Model Description: 2x2 crossover
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- SCD-101 (Experimental): SCD-101 dosed TID for 28-days
  Interventions: Drug: SCD-101
- Placebo (Placebo Comparator): Placebo dosed TID for 28-days
  Interventions: Drug: SCD-101

INTERVENTIONS:
Drug: SCD-101 — Administered as gelatin capsules

SUMMARY:
The purpose of this study is to determine the safety and clinical effects of SCD-101 when given to adults with sickle cell disease.

DETAILED DESCRIPTION:
This is single site, dose- escalation study of SCD-101 in participants with homozygous sickle cell disease (S/S) or S/beta 0 Thalassemia. All participants will be monitored for safety, tolerability, and dose-limiting toxicities.

The study is divided into two parts. Part A is an open-label, non-randomized, non-placebo-controlled dose escalation study with a 28-day treatment phase and 14-day follow-up phase with five cohorts . Part B is a randomized, placebo-controlled, confirmatory 2x2 crossover cohort with a 28 day washout between periods, and a 28-day follow-up phase.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, 18-55 years of age
2. Homozygous sickle cell disease or S/beta 0 thalassemia
3. Hemoglobin F ≤10%
4. Hemoglobin ≥ 6.0 g/dL and ≤ 9.5 g/dL
5. Female participants of child bearing potential and male participants whose partner is a female of child bearing potential must be willing to use approved contraception during the trial and for 3 months following the end of treatment. Only barrier methods or complete abstinence are acceptable for this study. Participants using hormonal contraception (including morning-after-pill) and IUD are excluded unless willing/able to change to an acceptable form of contraception.
6. Ability to adhere to the study visit schedule and other protocol requirements
7. Ability to understand and the willingness to sign an informed consent document

Exclusion Criteria:

1. Red blood cell transfusion within 3 months of enrollment
2. Hydroxyurea treatment within 6 months of enrollment
3. Painful or other acute sickle cell event that required a hospitalization within 4-weeks of enrollment
4. AST and/or ALT >3x upper limit of normal and/or creatinine >2x upper limit of normal or any other significant renal or hepatic impairment
5. Estimated creatinine clearance (CrCl) < 60 mL/min (Cockcroft- Gault formula) at screening.
6. QTc interval of >470 msec at trial entry and participant with congenital long QT syndrome.
7. No other significant sickle cell or non-sickle cell illness that would confound the results of the trial
8. Any condition that, in the view of the investigator, places the participant at risk because of participation in the trial, or may influence the result of the trial or the participant's ability to participate in the trial
9. Participant pregnant or nursing an infant or planning pregnancy during the course of the trial
10. History of allergic reactions attributed to sorghum or compounds of similar chemical or biologic composition (such as Nicosan, Niprisan, Jobelyn or Xickle).
11. Other investigational drug use within 3 months of enrollment
12. PROMIS Fatigue Questionnaire 8a T-score ˂ 44.3

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2015-02 (Actual); Primary Completion 2023-11 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Determine the safety, tolerability, and dose limiting toxicities of escalating doses of SCD-101, assessed by frequency and severity of adverse events (AEs), and changes in vital signs, 12-lead ECGs and laboratory assessments as compared to baseline | From the time the participant is administered the first dose through the final follow-up (18 weeks)

SECONDARY OUTCOMES:
Determine the effect of escalating doses of SCD-101 on the mean change in hemoglobin form base line | From the time the participant is accessed at baseline through the final follow-up (18 weeks)
Determine the effect of escalating doses of SCD-101 on the mean change in percent reticulocytes from baseline | From the time the participant is accessed at baseline through the final follow-up (18 weeks)
Determine the effect of escalating doses of SCD-101 on the mean change from baseline in red blood cell hemolysis as measured by lactate dehydrogenase (LDH) and indirect bilirubin. | From the time the participant is accessed at baseline through the final follow-up (18 weeks)
Determine the effect of escalating doses of SCD-101 on the mean change from baseline in fatigue as measured by the PROMIS fatigue questionnaire | From the time the participant is accessed at baseline through the final follow-up (18 weeks)
Determine the effect of escalating doses of SCD-101 on the mean change from baseline in the percent of venous circulating sickle red blood cells | From the time the participant is accessed at baseline through the final follow-up (18 weeks)
Determine the effect of escalating doses of SCD-101 on the mean change from baseline in functional capacity as measured by the 6-Minute Walk Test | From the time the participant is accessed at baseline through the final follow-up (18 weeks)

OTHER OUTCOMES:
Part B: Exploratory Outcome Measure the mean change from baseline in sleep interference as measured by the PROMIS sleep interference questionnaire | From the time the participant is accessed at baseline through the final follow-up (18 weeks)
Part B: Exploratory Outcome Measure the mean change from baseline in pain interference as measured by the PROMIS pain interference questionnaire | From the time the participant is accessed at baseline through the final follow-up (18 weeks)
Part B: Exploratory Outcome Measure the mean change from baseline in patient reported daily pain as measured by a Numeric Rating Scale (NRS 0-10) | From the time the participant is accessed at baseline through the final follow-up (18 weeks)
Part B: Exploratory Outcome Measure the mean change from baseline in analgesic usage as measured by patient medication diary | From the time the participant is accessed at baseline through the final follow-up (18 weeks)
Part B: Exploratory Outcome Measure the mean:change from baseline in exercise and sleep activity as measured by wrist actigraphy | From the time the participant is accessed at baseline through the final follow-up (18 weeks)
Part B: Exploratory Outcome Measure the mean:change from baseline in plasma inflammatory cytokines as measured by ELISA | From the time the participant is accessed at baseline through the final follow-up (18 weeks)

CONTACTS AND LOCATIONS:
Overall Officials: John Muthu, MD, Principal Investigator — King's County Hospital
Locations (1):
- King's County Hospital, Brooklyn, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wambebe C, Khamofu H, Momoh JA, Ekpeyong M, Audu BS, Njoku OS, Bamgboye EA, Nasipuri RN, Kunle OO, Okogun JI, Enwerem MN, Audam JG, Gamaniel KS, Obodozie OO, Samuel B, Fojule G, Ogunyale O. Double-blind, placebo-controlled, randomised cross-over clinical trial of NIPRISAN in patients with Sickle Cell Disorder. Phytomedicine. 2001 Jul;8(4):252-61. doi: 10.1078/0944-7113-00040. PMID 11515714
- [Background] Iyamu EW, Turner EA, Asakura T. In vitro effects of NIPRISAN (Nix-0699): a naturally occurring, potent antisickling agent. Br J Haematol. 2002 Jul;118(1):337-43. doi: 10.1046/j.1365-2141.2002.03593.x. PMID 12100171
- [Background] Iyamu EW, Turner EA, Asakura T. Niprisan (Nix-0699) improves the survival rates of transgenic sickle cell mice under acute severe hypoxic conditions. Br J Haematol. 2003 Sep;122(6):1001-8. doi: 10.1046/j.1365-2141.2003.04536.x. PMID 12956772
- [Background] Swift, RA, Nathan, S, Tripathi, P, Chen, Q, Asakura,T (2009, September). Research Preview on Improving Nicosan™/Xickle™: A Phyto-Medicine for the Treatment of Sickle Cell Disease. Paper presented at the meeting of the Sickle Cell Disease Association of America, Orlando, FL.
- [Derived] Li Q, Henry ER, Hofrichter J, Smith JF, Cellmer T, Dunkelberger EB, Metaferia BB, Jones-Straehle S, Boutom S, Christoph GW, Wakefield TH, Link ME, Staton D, Vass ER, Miller JL, Hsieh MM, Tisdale JF, Eaton WA. Kinetic assay shows that increasing red cell volume could be a treatment for sickle cell disease. Proc Natl Acad Sci U S A. 2017 Jan 31;114(5):E689-E696. doi: 10.1073/pnas.1619054114. Epub 2017 Jan 17. PMID 28096387